CLINICAL TRIAL: NCT05310474
Title: Does an Active Range of Motion Monitor Improve Outcomes and Decrease Cost for Patients Undergoing Total Knee Arthroplasty?
Brief Title: Does an Active Range of Motion Monitor Improve Outcomes/Decrease Cost for Patients Undergoing Total Knee Arthroplasty?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Force Therapeutics (Industry)
Collaborators: OSI Orthopedics and Sports Medicine (Unknown); Rehab 360 Knee Glider (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Rehab360 Knee Glider
Record Dates: First submitted 2021-12-14; First posted 2022-04-05 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Total Knee Arthroplasty (TKA)

STUDY DESIGN:
Intervention Model Description: This study includes 3 arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (No Intervention): Upon consent, patients will be randomized to receive standard of care, and not be given the active range of motion monitor (the knee glider) two weeks prior to surgery. All patients enrolled in the study will have access to Force Therapeutics, patient engagement and outcome collection system utilized by OSI Orthopedic & Sports Medicine.
- Group B (Experimental): Upon consent, patients will be randomized to receive the active range of motion monitor (the knee glider) close to surgery to use postoperatively (through week 4). All patients enrolled in the study will have access to Force Therapeutics, patient engagement and outcome collection system utilized by OSI Orthopedic & Sports Medicine.
  Interventions: Device: Knee Glider
- Group A (Experimental): Upon consent, patients will be randomized to receive the active range of motion monitor (the knee glider) Receives Knee Glider 2 weeks prior to surgery to utilize through postoperative week 4. All patients enrolled in the study will have access to Force Therapeutics, patient engagement and outcome collection system utilized by OSI Orthopedic & Sports Medicine.
  Interventions: Device: Knee Glider

INTERVENTIONS:
Device: Knee Glider — The purpose of this study is to study the efficacy of a remote range of motion monitor, the Knee Glider, alongside a patient engagement platform, Force Therapeutics, on clinical improvements and cost following primary TKA.
  Arms: Group A; Group B

SUMMARY:
The purpose of this study is to study the efficacy of a remote range of motion monitor, the Knee Glider, alongside a patient engagement platform, Force Therapeutics, on clinical improvements and cost following primary TKA.

DETAILED DESCRIPTION:
The purpose of this study is to study the efficacy of a remote range of motion monitor, the Knee Glider, alongside a patient engagement platform, Force Therapeutics, on clinical improvements and cost following primary TKA. Patients will be given the opportunity to participate, and enrolled and consented participants will be treated and followed by physicians from OSI Orthopedic & Sports Medicine. Upon consent, patients will be randomized to receive the active range of motion monitor (the knee glider) two weeks prior to surgery, near day of surgery to use postoperatively, or standard of care (no knee glider). All patients enrolled in the study will have access to Force Therapeutics, patient engagement and outcome collection system utilized by OSI Orthopedic & Sports Medicine. Enrolled subjects will be followed from the time of consent, through 6 months following surgery. Patients who are randomized into groups receiving the knee glider will receive the knee glider for up to 4 weeks following surgery, and compliance will be monitored. The hypothesis of this study is that patients who utilize an active range of motion monitor (the knee glider) will have improved clinical outcomes over patients receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone Total Knee Arthroplasty (TKA) and have agreed to participate in this study.

Exclusion Criteria:

* Individuals who have not undergone TKA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Patient Characteristics | Baseline
  Intended to collect patient demographics, contact information, birth date, surgery date, age and other baseline demographic variables.
Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) | Baseline, 2 Weeks Post Op, 6 Weeks Post Op, 12 Weeks Post Op, 6 Months Post Op,
  Intended to elicit people's opinions about the difficulties they experience due to problems with their knee and covers aspects of pain, functional limitations and knee-related quality of life.
  KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) | 6 Weeks Post Op
  Intended to elicit people's opinions about the difficulties they experience due to problems with their knee and covers aspects of pain, functional limitations and knee-related quality of life.
  KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) | 12 Weeks Post Op
  Intended to elicit people's opinions about the difficulties they experience due to problems with their knee and covers aspects of pain, functional limitations and knee-related quality of life.
  KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) | 6 Months Post Op
  Intended to elicit people's opinions about the difficulties they experience due to problems with their knee and covers aspects of pain, functional limitations and knee-related quality of life.
  KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline
  1. The WOMAC is a disease-specific tool used for people with hip or knee OA to measure physical function, pain, and stiffness in the past 48 hours.
  2. The WOMAC is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items).
  3. Scores can be calculated for each subscale and a total score is calculated by adding all 3 subscale scores. Higher points signify higher levels of functional difficulty.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 Weeks Post Op
  1. The WOMAC is a disease-specific tool used for people with hip or knee OA to measure physical function, pain, and stiffness in the past 48 hours.
  2. The WOMAC is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items).
  3. Scores can be calculated for each subscale and a total score is calculated by adding all 3 subscale scores. Higher points signify higher levels of functional difficulty.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 Weeks Post Op
  1. The WOMAC is a disease-specific tool used for people with hip or knee OA to measure physical function, pain, and stiffness in the past 48 hours.
  2. The WOMAC is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items).
  3. Scores can be calculated for each subscale and a total score is calculated by adding all 3 subscale scores. Higher points signify higher levels of functional difficulty.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 Months Post Op
  1. The WOMAC is a disease-specific tool used for people with hip or knee OA to measure physical function, pain, and stiffness in the past 48 hours.
  2. The WOMAC is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items).
  3. Scores can be calculated for each subscale and a total score is calculated by adding all 3 subscale scores. Higher points signify higher levels of functional difficulty.
Veterans RAND 12 (VR-12) | Baseline
  a. The Veterans RAND 12 Item Health Survey (VR-12) is a patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Veterans RAND 12 (VR-12) | 6 Weeks Post Op
  The Veterans RAND 12 Item Health Survey (VR-12) is a patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Veterans RAND 12 (VR-12) | 12 Weeks Post Op
  The Veterans RAND 12 Item Health Survey (VR-12) is a patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Veterans RAND 12 (VR-12) | 6 Months Post Op
  The Veterans RAND 12 Item Health Survey (VR-12) is a patient-reported global health measure that is used to assess a patient's overall perspective of their health.
Force Patient Engagement | Baseline
  Engagement on the patient engagement platform including logins, exercise videos watched and patient recorded outcome measures (PROM) compliance during platform access
Force Patient Engagement | 2 Weeks Post Op
  Engagement on the patient engagement platform including logins, exercise videos watched and patient recorded outcome measures (PROM) compliance during platform access
Force Patient Engagement | 6 Weeks Post Op
  Engagement on the patient engagement platform including logins, exercise videos watched and patient recorded outcome measures (PROM) compliance during platform access
Force Patient Engagement | 12 Weeks Post Op
  Engagement on the patient engagement platform including logins, exercise videos watched and patient recorded outcome measures (PROM) compliance during platform access
Force Patient Engagement | 6 Months Post Op
  Engagement on the patient engagement platform including logins, exercise videos watched and patient recorded outcome measures (PROM) compliance during platform access
Range of Motion via the Knee Glider | Baseline
  Daily Knee Flexion and Extension for the duration of utilizing the knee glider
Range of Motion via the Knee Glider | 2 Weeks Post Op
  Daily Knee Flexion and Extension for the duration of utilizing the knee glider
Range of Motion via the Knee Glider | 6 Weeks Post Op
  Daily Knee Flexion and Extension for the duration of utilizing the knee glider
Range of Motion via the Knee Glider | 12 Weeks Post Op
  Daily Knee Flexion and Extension for the duration of utilizing the knee glider
Range of Motion (Exam / Patient Reported) | Baseline
  a. Knee Flexion and Extension via in clinic exam or patient reported via the Force Therapeutics Platform
Range of Motion (Exam / Patient Reported) | 2 Weeks Post Op
  a. Knee Flexion and Extension via in clinic exam or patient reported via the Force Therapeutics Platform (0 to 110 degrees)
Range of Motion (Exam / Patient Reported) | 6 Weeks Post Op
  a. Knee Flexion and Extension via in clinic exam or patient reported via the Force Therapeutics Platform (0 to 110 degrees)
Range of Motion (Exam / Patient Reported) | 12 Weeks Post Op
  a. Knee Flexion and Extension via in clinic exam or patient reported via the Force Therapeutics Platform (0 to 110 degrees)
Daily NRS Pain (Continuous) | Baseline
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain
Daily NRS Pain (Continuous) | 2 Weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain
Daily NRS Pain (Continuous) | 6 Weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain
Daily NRS Pain (Continuous) | 12 Weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain
Discharge Services Utilization & Cost | 6 Weeks Post Op
  The Discharge Services Utilization & Cost survey is intended collect patient discharge information. The survey consists of 16 questions asking about where they went for physical therapy, how much it costs, and if any adverse events resulted in admission to an Emergency Room or Urgent Care.
Discharge Services Utilization & Cost | 12 Weeks Post Op
  The Discharge Services Utilization & Cost survey is intended collect patient discharge information. The survey consists of 16 questions asking about where they went for physical therapy, how much it costs, and if any adverse events resulted in admission to an Emergency Room or Urgent Care.
Knee Glider Satisfaction | 2 Weeks Post Op
  The Knee Glider Satisfaction questionnaire is a 4 question survey asking about patient experience using the glider.
Knee Glider Satisfaction | 6 Weeks Post Op
  The Knee Glider Satisfaction questionnaire is a 4 question survey asking about patient experience using the glider.
Knee Glider Satisfaction | 12 Weeks Post Op
  The Knee Glider Satisfaction questionnaire is a 4 question survey asking about patient experience using the glider.
Total Joint Replacement (TJR) Satisfaction | 12 Weeks Post Op
  The TJR Satisfaction survey intends to understand patient experience and satisfaction results with their total joint replacement procedure.
Total Joint Replacement (TJR) Satisfaction | 6 Months Post Op
  The TJR Satisfaction survey intends to understand patient experience and satisfaction results with their total joint replacement procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Cornett, DO, Principal Investigator — OSI Orthopedic Sports Medicine